CLINICAL TRIAL: NCT05916677
Title: Virtual Reality-training in Theory of Mind in the Childhood Form of Myotonic Dystrophy Type 1
Acronym: TOM-VR-DM1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: TOM-VR-DM1
Record Dates: First submitted 2023-06-02; First posted 2023-06-23 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Myotonic Dystrophy Type 1
Keywords: Myotonic Dystrophy type 1; Theory of Mind; Virtual environment; Training protocol
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient remediate using the virtual training method (Experimental)
  Interventions: Other: Virtual Reality-training in Theory of Mind
- Patient remediate using the traditional training method (Active Comparator)
  Interventions: Other: Traditional training in Theory of Mind

INTERVENTIONS:
Other: Virtual Reality-training in Theory of Mind — Two social scenarios will be used in a virtual environement. Experimenter and subject participate in the scenario as friends of the main character, Nicolas. During the training session, experimenter asks structured questions about participant's awareness of a mental state. In the case of a wrong answer, a feedback-correction is provided via the avatar's thought bubbles. The participant has access to all avatars thought bubbles. In this way, he is able to compare the desires, beliefs or false beliefs of each story character.
  Participants included in this condition will also have an eye-tracking assessment before and after the training procedure.
  Arms: Patient remediate using the virtual training method
Other: Traditional training in Theory of Mind — The same two social scenarios are presented to the participant in a story-telling form. Participant has access to thought bubbles via an illustrated book. These trainings will take place in the same number of sessions and took place for a duration equivalent to those used in low immersion Virtual Reality mode. Each training session (EFB, BE, SOFB, ERA, FP, EFP) will be illustrated via visual aids taken from screenshots of the two virtual environments and the target protagonists.
  Arms: Patient remediate using the traditional training method

SUMMARY:
The ability of an individual to conceive some alternative representations and to behave in a flexible manner would emerge from preschool age and drastically improve between the ages of 3 and 5 (Doebel and Zelazo, 2013). They constitute, according to Diamond (2013), a prerequisite for the development of the Theory of Mind (ToM). Deficits in Executive Functions (EF) may therefore interfere with the child's ability to understand and adapt to social situations.

Treatment failures are often observed when traditional cognitive tools are used. This would be linked to the divergence between non-immersive tests and situations encountered in everyday life (Damasio, 1994; Priore Castelnuovo and Liccione, 2002). For this reason, an increasing number of researchers are using virtual reality for the rehabilitation of executive functions and Theory of Mind in patients with neurodevelopmental pathology (Millen, Edlin-White and Cobb, 2010) or brain damage (Le Gall, Besnard, Louisy, Richard and Allain 2008). There is currently no systematic evaluation of ToM in children with the infantile form of DM1 even though these abilities are considered particularly vulnerable and have a decisive impact on the subsequent development of interpersonal relationships.

This research will focus on studying the socio-emotional disorders associated with the infantile form of Myotonic Dystrophy type 1 (DM1). The axis that we propose to develop more specifically will be an interventional study with the aim of remediation with children from 5 to 16 years old suffering from the infantile form of DM1 via a training protocol in low-immersion Virtual Reality (VR) centered on emotional processing and theory of mind.

ELIGIBILITY:
Inclusion Criteria:

* 6 years and < 16 years of age
* Written informed consent
* Affiliate or beneficiary of a social security scheme
* Able to comply with all protocol requirements
* Infantile form of DM1 with molecular confirmation.
* Development without incident in the first year
* Normal development in the pre and neonatal period
* Native language French

Exclusion Criteria:

* Unable to participate in the study
* Inability to comply with protocol requirements
* Congenital form of DM1
* IQ<70 (Intellectual Disability)

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 95 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
NEPSY II | Through study completion, an average of 5 weeks
  Emotion Recognition and Standardized ToM

SECONDARY OUTCOMES:
WISC-V | Through study completion, on average 5 weeks
  Wechsler Scale is the international benchmark for measuring children's intelligence

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Psychologie, Boulogne-Billancourt, France